CLINICAL TRIAL: NCT01424670
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group Trial to Evaluate the Safety and Efficacy of Delamanid (OPC-67683) Administered Orally as 200 mg Total Daily Dose for Six Months in Patients With Pulmonary Sputum Culture-positive, Multidrug-resistant Tuberculosis
Brief Title: Safety and Efficacy Trial of Delamanid for 6 Months in Participants With Multidrug-resistant Tuberculosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 242-09-213
Record Dates: First submitted 2011-08-25; First posted 2011-08-29 (Estimated); Results first posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Multidrug-resistant Tuberculosis
Keywords: Multidrug-resistant tuberculosis
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant | interventions — OPC-67683

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Delamanid + OBR (Experimental): In the first period of this study, known as the 6-month Intensive Period, participants were randomized to receive 100 mg delamanid orally BID (morning and evening) + OBR for 2 months, followed by 200 mg delamanid QD (every morning) + OBR for 4 months.
  Following the 6-month Intensive Period, participants entered the second period of the study, known as the Continuation Period, wherein OBR was administered alone for 12 to 18 months.
  OBR given throughout the study was administered as per WHO guidelines and national treatment norms.
  Interventions: Drug: Delamanid + OBR
- Placebo + OBR (Placebo Comparator): In the first period of this study, known as the 6-month Intensive Period, participants were randomized to receive placebo orally BID (morning and evening) + OBR for 2 months followed by placebo QD (every morning) + OBR for 4 months.
  Following the 6-month Intensive Period, participants entered the second period of the study, known as the Continuation Period, wherein OBR was administered alone for 12 to 18 months.
  OBR given throughout the study was administered as per WHO guidelines and national treatment norms.
  Interventions: Drug: Placebo + OBR

INTERVENTIONS:
Drug: Delamanid + OBR — The assigned doses of delamanid were administered with an OBR. The selection and administration of the OBR were based on WHO's guidelines for the programmatic management of drug-resistant TB, in conjunction with national TB program guidelines in each country.
  Arms: Delamanid + OBR
Drug: Placebo + OBR — Matching placebo was administered with an OBR. The selection and administration of the OBR were based on WHO's guidelines for the programmatic management of drug-resistant TB, in conjunction with national TB program guidelines in each country.
  Arms: Placebo + OBR

SUMMARY:
The purpose of this trial is to determine whether delamanid is effective in the treatment of multidrug-resistant tuberculosis (MDR TB) in combination with other MDR TB medications during 6 months of treatment.

DETAILED DESCRIPTION:
The primary objective of this trial is to evaluate the efficacy of delamanid administered orally as 100 milligrams (mg) twice daily (BID) for 2 months followed by 200 mg once daily (QD) for 4 months in combination with an optimized background treatment regimen (OBR) versus placebo with OBR during the 6-month Intensive Period of MDR TB treatment. Following the 6-month Intensive Period, OBR was administered alone during the Continuation Period for 12 to 18 months (from Month 7 up to Month 24). The trial also included a post-treatment follow-up period of 6 to 12 months (Month 19 to Month 24 to the end of Month 30). OBR given throughout the study was administered as per World Health Organization (WHO) guidelines and national treatment norms.

This trial is a multicenter, randomized, double-blind, stratified, placebo-controlled trial that was conducted globally in 2 parallel groups at 17 sites in 7 countries qualified to treat MDR TB.

ELIGIBILITY:
Inclusion Criteria:

* Provide written, informed consent
* Current diagnosis of MDR TB
* Chest radiograph consistent with TB
* Able to produce sputum
* Negative urine pregnancy test and agree to use a highly effective method of birth control and/or adequate method of contraception

Exclusion Criteria:

* Allergy to any nitro-imidazoles or nitro-imidazole derivates
* Diseases or conditions in which the use of nitro-imidazoles or nitro-imidazole derivates is contra-indicated
* Use of disallowed medications
* Renal impairment
* Abnormal electrocardiogram (ECG) results
* Cardiovascular disorders
* Body mass index (BMI) < 16 kg/m^2
* Karnofsky score < 50%
* Significant metabolic, gastrointestinal, neurological, psychiatric, or endocrine diseases, active malignancy
* Alcohol abuse
* Pregnant, breast-feeding, or planning to conceive or father a child
* Recent use of methadone, benzodiazepines, cocaine, amphetamine/methamphetamine, tetrahydrocannabinol, barbiturates, and opiates
* Previous exposure to delamanid
* Administered an investigational medicinal product (IMP) within 1 month prior to Screening (Days -21 to -2).
* Evidence of extensively drug-resistant TB based on the definition from WHO
* Human immunodeficiency virus (HIV) co-infection for participants screened at sites not participating in the HIV subtrial (data from the HIV subtrial will be reported separately from the Clinical Study Report for Study 242-09-213).

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2011-09-02 (Actual); Primary Completion 2016-07-04 (Actual); Study Completion 2016-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Development, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (17):
- Tartu, Estonia
- Riga, Latvia
- Lithuania (2):
  - Šiauliai
  - Vilnius
- Moldova (2):
  - Chisinau
  - Vorniceni
- Peru (4):
  - Alfonso Ugarte
  - Comas
  - El Agustino
  - Lima Cercado
- Philippines (4):
  - Dasmariñas, Cavite
  - Quezon City, National Capital Region
  - Makati City
  - Quezon City
- South Africa (3):
  - Cape Town
  - Durban
  - Klerksdorp

REFERENCES:
- [Derived] von Groote-Bidlingmaier F, Patientia R, Sanchez E, Balanag V Jr, Ticona E, Segura P, Cadena E, Yu C, Cirule A, Lizarbe V, Davidaviciene E, Domente L, Variava E, Caoili J, Danilovits M, Bielskiene V, Staples S, Hittel N, Petersen C, Wells C, Hafkin J, Geiter LJ, Gupta R. Efficacy and safety of delamanid in combination with an optimised background regimen for treatment of multidrug-resistant tuberculosis: a multicentre, randomised, double-blind, placebo-controlled, parallel group phase 3 trial. Lancet Respir Med. 2019 Mar;7(3):249-259. doi: 10.1016/S2213-2600(18)30426-0. Epub 2019 Jan 7. PMID 30630778

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 511 participants were randomized to receive investigational medicinal product (IMP) and an optimized background treatment regimen (OBR) for 6 months, followed by OBR treatment alone for 12-18 months. The trial also included a post-treatment follow-up period of 6-12 months. Participants who stopped taking IMP and/or OBR could remain in the study.
Groups:
- Delamanid + OBR: In the first period of this study, known as the 6-month Intensive Period, participants were randomized to receive 100 milligrams (mg) delamanid orally twice daily (BID) (morning and evening) + OBR for 2 months, followed by 200 mg delamanid once daily (QD) (every morning) + OBR for 4 months.
  Following the 6-month Intensive Period, participants entered the second period of the study, known as the Continuation Period, wherein OBR was administered alone for 12 to 18 months.
- Placebo + OBR: In the first period of this study, known as the 6-month Intensive Period, participants were randomized to receive placebo orally BID (morning and evening) + OBR for 2 months followed by placebo QD (every morning) + OBR for 4 months.
  Following the 6-month Intensive Period, participants entered the second period of the study, known as the Continuation Period, wherein OBR was administered alone for 12 to 18 months.
Period: 6-Month Intensive Period (182 Days)
Arm/Group | Delamanid + OBR | Placebo + OBR
Started | 341 | 170
Received at Least 1 Dose of Study Drug | 341 | 170
Completed (The duration of the 6-month Intensive Period was over 182 days from the date of the first dose.) | 322 | 156
Not Completed | 19 | 14
Not completed — Adverse Event | 2 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Met Protocol Withdrawal Criteria | 2 | 1
Not completed — Physician Decision | 2 | 3
Not completed — Withdrawal by Subject | 13 | 7
Period: Continuation Period
Arm/Group | Delamanid + OBR | Placebo + OBR
Started | 322 | 156
Completed | 288 | 142
Not Completed | 34 | 14
Not completed — Adverse Event | 13 | 5
Not completed — Lost to Follow-up | 2 | 0
Not completed — Met Protocol Withdrawal Criteria | 1 | 1
Not completed — Physician Decision | 5 | 4
Not completed — Withdrawal by Subject | 13 | 4

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat Sample comprised all participants who were randomized to receive either delamanid + OBR or placebo + OBR in this study.
Groups:
- Delamanid + OBR: In the first period of this study, known as the 6-month Intensive Period, participants were randomized to receive 100 mg delamanid orally BID (morning and evening) + OBR for 2 months, followed by 200 mg delamanid QD (every morning) + OBR for 4 months.
  Following the 6-month Intensive Period, participants entered the second period of the study, known as the Continuation Period, wherein OBR was administered alone for 12 to 18 months.
- Total: Total of all reporting groups
Arm/Group | Delamanid + OBR | Placebo + OBR | Total
Number analyzed (Participants) | 341 | 170 | 511
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.3 (12.1) | 34.4 (12.2) | 34.3 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 45 | 143
  Male | 243 | 125 | 368

OUTCOME MEASURES:

1. Primary Outcome: Time To Sputum Culture Conversion (SCC) During 6-Month Intensive Period Using The Mycobacteria Growth Indicator Tube (MGIT) System
Description: SCC at 6 months was determined by the observation of a sputum specimen negative for growth of mycobacterium tuberculosis (MTB) using the MGIT culture system, followed by at least 1 confirmatory negative sputum culture at least 25 days after the first negative and not followed by a confirmed positive (defined as at least 2 observed positive results, not taking into account indeterminate, missing, or contaminated results). 2 specimens were collected at each visit and an algorithm in the statistical analysis plan (SAP) was used to define a single representative result. Time to SCC was then defined as the interval between the date of first dose of IMP and the date of first of 2 consecutive negative single representative time points that were at least 25 days apart. The median time in days to SCC up to Month 6 is presented.
Time Frame: Month 6
Population: The modified intent-to-treat (MITT) sample comprised all randomized participants who had a positive sputum culture for MTB in MGIT and were resistant to both isoniazid and rifampicin from the sputum samples collected on either Day -1 or Day 1, or both.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Delamanid + OBR: In the 6-month Intensive Period, participants were randomized to receive 100 mg delamanid orally BID (morning and evening) + OBR for 2 months, followed by 200 mg delamanid QD (every morning) + OBR for 4 months.
- Placebo + OBR: In the 6-month Intensive Period, participants were randomized to receive placebo orally BID (morning and evening) + OBR for 2 months followed by placebo QD (every morning) + OBR for 4 months.
Arm/Group | Delamanid + OBR | Placebo + OBR
Number analyzed (Participants) | 226 | 101
Days | 51 [43 to 57] | 57 [56 to 64]
Statistical Analysis 1: Comparison: Delamanid + OBR vs Placebo + OBR; Comparison of distributions of time to SCC using the MGIT culture system during the 6-month (26-week) Intensive Period; Test type: Superiority; p = 0.0562, Modified Peto-Peto test — For testing the null hypothesis, the distribution of the time to SCC within the 6-month Intensive Period were compared between the 2 treatment groups using the stratified modified Peto-Peto modification of Gehan's Wilcoxon rank sum test

2. Secondary Outcome: Proportion of Participants With SCC At 2 And 6 Months Using MGIT
Description: SCC was evaluated at 2 and 6 months (6-month Intensive Period) using MGIT. SCC at 2 months was defined to occur at the date of collection of the first sputum specimen with mycobacterial culture negative for growth of MTB using MGIT culture, followed by at least 1 confirmatory negative MGIT culture result at least 25 days after the first negative specimen and not followed by any sputum specimens positive for growth in the MGIT culture at any point up to 3 months (Week 12).
  SCC at 6 months was determined by the observation of a sputum specimen negative for growth of MTB using the MGIT culture system, followed by at least 1 confirmatory negative sputum culture at least 25 days after the first negative and not followed by a confirmed positive (defined as at least 2 observed positive results, not taking into account indeterminate, missing, or contaminated results). 2 specimens were collected at each visit and an algorithm in the SAP was used to define a single representative result.
Time Frame: Month 2 and Month 6
Population: The MITT sample comprised all randomized participants who had a positive sputum culture for MTB in MGIT and were resistant to both isoniazid and rifampicin from the sputum samples collected on either Day -1 or Day 1, or both.
Measure: Count of Participants; unit: Participants
Arm/Group | Delamanid + OBR | Placebo + OBR
Number analyzed (Participants) | 226 | 101
Participants
  At Month 2 | 132 | 54
  At Month 6 | 198 | 87
Statistical Analysis 1: Comparison: Delamanid + OBR vs Placebo + OBR; Statistical comparison of proportion of participants with SCC at 2 months; Test type: Superiority — For testing the homogeneity of proportions, 2 samples were compared using the stratified Cochran-Mantel-Haenszel test; p = 0.3818, Cochran-Mantel-Haenszel; Ratio of Probability = 1.096, 95% CI 2-sided [0.889 to 1.352] — The stratified Cochran-Mantel-Haenszel test statistics were used for estimation
Statistical Analysis 2: Comparison: Delamanid + OBR vs Placebo + OBR; Statistical comparison of proportion of participants with SCC at 6 months; Test type: Superiority — For testing the homogeneity of proportions, 2 samples were compared using the stratified Cochran-Mantel-Haenszel test; p = 0.7131, Cochran-Mantel-Haenszel; Ratio of Probability = 1.017, 95% CI 2-sided [0.927 to 1.115] — The stratified Cochran-Mantel-Haenszel test statistics were used for estimation

3. Secondary Outcome: Proportion of Participants With Sustained SCC At Month 18, Month 24, And Month 30 Using MGIT
Description: Sustained SCC was defined as SCC achieved by Month 6 and not followed by a confirmed positive thereafter, where confirmed positive was defined as 2 or more observed positive single representative culture results, not taking into account indeterminate, missing, or contaminated results. Sustained SCC was analyzed at Month 18 to 30 using MGIT.
Time Frame: Month 18, Month 24, and Month 30
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Delamanid + OBR | Placebo + OBR
Number analyzed (Participants) | 226 | 101
Participants
  At 18 months | 180 | 83
  At 24 months | 178 | 82
  At 30 months | 173 | 78
Statistical Analysis 1: Comparison: Delamanid + OBR vs Placebo + OBR; Statistical comparison of proportion with sustained SCC at Month 18; Test type: Superiority; p = 0.5945, Cochran-Mantel-Haenszel; Relative Ratio of Probability = 0.969, 95% CI 2-sided [0.866 to 1.084]
Statistical Analysis 2: Comparison: Delamanid + OBR vs Placebo + OBR; Statistical comparison of proportion with sustained SCC at Month 24; Test type: Superiority; p = 0.6164, Cochran-Mantel-Haenszel; Relative Ratio of Probability = 0.97, 95% CI 2-sided [0.864 to 1.089]
Statistical Analysis 3: Comparison: Delamanid + OBR vs Placebo + OBR; Statistical comparison of proportion with sustained SCC at Month 30; Test type: Superiority; p = 0.8951, Cochran-Mantel-Haenszel; Relative Ratio of Probability = 0.991, 95% CI 2-sided [0.872 to 1.127]

4. Secondary Outcome: Treatment Outcomes Assessed By Principal Investigators (PI)At The End Of Treatment With OBR
Description: Final treatment outcomes were assessed by the Principal Investigator (PI) at the end of treatment with OBR (24 months post randomization) according to the 2008 World Health Organization (WHO) outcome definitions for treating participants with multidrug-resistant tuberculosis (MDR TB). Frequency counts and percentage of participants achieving favorable and unfavorable outcomes were provided by treatment group. Participants who had non-missing Principal Investigator assessed treatment outcomes at the end of treatment with OBR were included in the analysis.
Time Frame: Month 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Delamanid + OBR | Placebo + OBR
Number analyzed (Participants) | 226 | 101
Participants
  Favorable outcome | 182 | 85
  Unfavorable outcome | 42 | 16
  Missing PI Assessments | 2 | 0
Statistical Analysis 1: Comparison: Delamanid + OBR vs Placebo + OBR; Statistical comparison of proportions with favorable treatment outcomes assessed by the Principal Investigator; Test type: Superiority; p = 0.5269, Cochran-Mantel-Haenszel; Relative Ratio of Probability = 0.965, 95% CI 2-sided [0.869 to 1.073]

5. Secondary Outcome: Number of Participants Who Developed Resistance To Delamanid
Description: Acquired resistance was defined as a post-baseline resistant result at any time point after a Baseline susceptible result. The overall resistance to delamanid during the trial was assessed.
Time Frame: Up to Month 30
Population: The intent-to-treat (ITT) sample comprised all randomized participants.
Measure: Number; unit: participants
Arm/Group | Delamanid + OBR | Placebo + OBR
Number analyzed (Participants) | 341 | 170
participants | 3 | 0

6. Secondary Outcome: Mean (Time Averaged) Area Under The Curve (AUC) Of Change From Baseline In Time To Detection (TTD) To Month 6 Using MGIT
Description: The value for TTD was defined (in days) as the time interval from inoculation until a MGIT machine detects a positive signal for a sputum culture. The AUC of the change from Baseline for TTD in days (from Baseline to Month 6) summarizes the overall participant response for the treatment period. The change from Baseline in original time to detection of MGIT positive signal, in days, up to 6 months was performed using AUC in MGIT. The Baseline was defined as the average of Day -1 and Day 1 values if cultures on both days were positive; if only 1 culture was positive, the value for TTD for the positive culture was used as the Baseline.
  The TTD is Time to Detection measured by day, so the unit of AUC of change from baseline in TTD is day*day. Since "Mean AUC" is reported, which is actually "Time Averaged AUC," the AUC was divided by the duration of the observation, and thus the unit of the Mean AUC is day.
Time Frame: Baseline, up to Month 6
Population: The MITT sample comprised all randomized participants who had a positive sputum culture for MTB in MGIT and were resistant to both isoniazid and rifampicin from the sputum samples collected on either Day -1 or Day 1, or both, who had both a baseline and at least one post baseline TTD value.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Delamanid + OBR | Placebo + OBR
Number analyzed (Participants) | 221 | 98
days | 21.9 (9.44) | 23.3 (8.93)
Statistical Analysis 1: Comparison: Delamanid + OBR vs Placebo + OBR; Statistical comparison of mean AUC of change from Baseline; Test type: Superiority; p = 0.6986, ANCOVA; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.9 to 1.3]

7. Secondary Outcome: Mean Change From Baseline In TTD Using The MGIT System
Description: The value for TTD was defined (in days) as the time interval from inoculation until a MGIT machine detects a positive signal for a sputum culture during the routine 42-day incubation period. TTD analysis was based only on the corresponding qualitative sputum results of pure positive and pure negative cultures in days and hours of the initial positive signal for a culture from the MGIT printout. Mean change is reported for Baseline, Week 1, Week 2, Week 3, Week 24, Week 26, and Last visit (Month 18 or last visit for participants treated beyond Month 18).
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 24, Week 26, and Last visit (Month 18 or last visit for participants treated beyond Month 18)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Delamanid + OBR | Placebo + OBR
Number analyzed (Participants) | 226 | 101
days
  At Baseline: number analyzed (Participants) | 222 | 98
  At Baseline | 16.7 (7.9) | 15.4 (7.7)
  At Week 1: number analyzed (Participants) | 204 | 94
  At Week 1 | 20.8 (10.3) | 19.9 (11.1)
  Change from Baseline at Week 1: number analyzed (Participants) | 204 | 94
  Change from Baseline at Week 1 | 4.3 (7.9) | 4.8 (7.8)
  At Week 2: number analyzed (Participants) | 206 | 87
  At Week 2 | 24.6 (11.5) | 23.1 (11.4)
  Change from Baseline at Week 2: number analyzed (Participants) | 206 | 87
  Change from Baseline at Week 2 | 7.7 (8.9) | 7.5 (7.8)
  At Week 3: number analyzed (Participants) | 209 | 89
  At Week 3 | 28.4 (11.8) | 25.5 (12.4)
  Change from Baseline at Week 3: number analyzed (Participants) | 209 | 89
  Change from Baseline at Week 3 | 11.6 (9.8) | 10.4 (9.6)
  At Week 24: number analyzed (Participants) | 195 | 80
  At Week 24 | 40.4 (6.6) | 41.3 (3.9)
  Change from Baseline at Week 24: number analyzed (Participants) | 195 | 80
  Change from Baseline at Week 24 | 23.4 (10.2) | 25.5 (8.3)
  At Week 26: number analyzed (Participants) | 188 | 82
  At Week 26 | 40.6 (5.9) | 40.5 (5.5)
  Change from Baseline at Week 26: number analyzed (Participants) | 188 | 82
  Change from Baseline at Week 26 | 23.8 (9.5) | 24.6 (9.4)
  At Last Visit: number analyzed (Participants) | 222 | 98
  At Last Visit | 39.4 (8.4) | 40.3 (6.3)
  Change from Baseline at Last Visit: number analyzed (Participants) | 222 | 98
  Change from Baseline at Last Visit | 22.7 (10.7) | 24.9 (9.5)
Statistical Analysis 1: Comparison: Delamanid + OBR vs Placebo + OBR; Statistical analysis for Week 1; Test type: Superiority; p = 0.6825, ANCOVA
Statistical Analysis 2: Comparison: Delamanid + OBR vs Placebo + OBR; Statistical analysis for Week 2; Test type: Superiority; p = 0.807, ANCOVA
Statistical Analysis 3: Comparison: Delamanid + OBR vs Placebo + OBR; Statistical analysis for Week 3; Test type: Superiority; p = 0.269, ANCOVA
Statistical Analysis 4: Comparison: Delamanid + OBR vs Placebo + OBR; Statistical analysis for Week 24; Test type: Superiority; p = 0.2333, ANCOVA
Statistical Analysis 5: Comparison: Delamanid + OBR vs Placebo + OBR; Statistical analysis for Month 6; Test type: Superiority; p = 0.9397, ANCOVA

8. Secondary Outcome: Proportion of Participants With Final Outcome At Month 30 As A Treatment Success Or Failure (Including Relapse) Using MGIT
Description: Treatment success was defined as achieving SCC by 6 months using MGIT, completing the trial out to 30 months with sustained SCC and alive at the last contact for follow-up. All other participants were treatment failures who failed to achieve SCC by Month 6, achieved SCC but have a confirmed positive, early terminate from the trial prior to the Month 30 visit but are alive at the last contact for follow-up, lost to follow-up and vital status unknown and death.
Time Frame: Month 30
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Delamanid + OBR | Placebo + OBR
Number analyzed (Participants) | 226 | 101
Participants
  Success | 173 | 78
  Failure | 53 | 23
Statistical Analysis 1: Comparison: Delamanid + OBR vs Placebo + OBR; Statistical comparison of proportion with treatment success at Month 30; Test type: Superiority; p = 0.8951, Cochran-Mantel-Haenszel; Relative Ratio of Probability = 0.991, 95% CI 2-sided [0.872 to 1.127]

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the study (30 months)
Description: Adverse events were collected for randomized participants who received any amount of study drug, regardless of any protocol deviation or violation.
Arm/Group | Delamanid + OBR | Placebo + OBR
All-Cause Mortality (participants affected / at risk) | 18/341 | 8/170
Serious Adverse Events (participants affected / at risk) | 89/341 | 47/170
Other Adverse Events (participants affected / at risk) | 335/341 | 165/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Delamanid + OBR (N=341) | Placebo + OBR (N=170)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 | 0
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0
Cor pulmonale (Cardiac disorders) | 1 | 0
Metabolic cardiomyopathy (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 1 | 1
Deafness bilateral (Ear and labyrinth disorders) | 4 | 4
Goitre (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Glaucoma (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0
Gastroduodenitis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Ileal perforation (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Oedematous pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 2 | 0
Hypothermia (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Hepatitis alcoholic (Hepatobiliary disorders) | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 2 | 0
Hepatotoxicity (Hepatobiliary disorders) | 3 | 2
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 1 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 2
Appendicitis perforated (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 1
Lung abscess (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 2
Pneumonia necrotising (Infections and infestations) | 0 | 1
Pneumonia viral (Infections and infestations) | 1 | 0
Pulmonary tuberculoma (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 2 | 1
Sepsis (Infections and infestations) | 1 | 1
Tuberculoma of central nervous system (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 11 | 3
Tuberculous pleurisy (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 2 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 2
Chest injury (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
Kidney contusion (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 6 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 3
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Acute psychosis (Psychiatric disorders) | 2 | 0
Alcohol abuse (Psychiatric disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Anxiety disorder (Psychiatric disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 1
Delirium tremens (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 1 | 1
Major depression (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 3 | 1
Reactive psychosis (Psychiatric disorders) | 1 | 0
Substance-induced psychotic disorder (Psychiatric disorders) | 2 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 5
Azotaemia (Renal and urinary disorders) | 0 | 2
Nephropathy toxic (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bullous lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary haematoma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 2
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Delamanid + OBR (N=341) | Placebo + OBR (N=170)
Anaemia (Blood and lymphatic system disorders) | 17 | 9
Palpitations (Cardiac disorders) | 19 | 12
Deafness bilateral (Ear and labyrinth disorders) | 15 | 9
Hypoacusis (Ear and labyrinth disorders) | 15 | 15
Tinnitus (Ear and labyrinth disorders) | 71 | 36
Vision blurred (Eye disorders) | 13 | 10
Abdominal pain (Gastrointestinal disorders) | 33 | 21
Abdominal pain upper (Gastrointestinal disorders) | 35 | 28
Constipation (Gastrointestinal disorders) | 12 | 13
Diarrhoea (Gastrointestinal disorders) | 62 | 33
Dyspepsia (Gastrointestinal disorders) | 33 | 14
Gastritis (Gastrointestinal disorders) | 76 | 27
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 19 | 11
Nausea (Gastrointestinal disorders) | 95 | 56
Toothache (Gastrointestinal disorders) | 29 | 17
Vomiting (Gastrointestinal disorders) | 92 | 39
Asthenia (General disorders) | 27 | 10
Chest pain (General disorders) | 22 | 8
Injection site pain (General disorders) | 24 | 20
Hepatotoxicity (Hepatobiliary disorders) | 20 | 11
Bronchitis (Infections and infestations) | 19 | 13
Influenza (Infections and infestations) | 21 | 6
Nasopharyngitis (Infections and infestations) | 71 | 43
Pharyngitis (Infections and infestations) | 32 | 23
Rhinitis (Infections and infestations) | 13 | 10
Upper respiratory tract infection (Infections and infestations) | 49 | 21
Urinary tract infection (Infections and infestations) | 36 | 15
Contusion (Injury, poisoning and procedural complications) | 22 | 10
Decreased appetite (Metabolism and nutrition disorders) | 26 | 9
Hyperuricaemia (Metabolism and nutrition disorders) | 34 | 22
Hypokalaemia (Metabolism and nutrition disorders) | 53 | 29
Hypomagnesaemia (Metabolism and nutrition disorders) | 20 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 116 | 65
Back pain (Musculoskeletal and connective tissue disorders) | 44 | 31
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 21 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 31 | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 24 | 16
Dizziness (Nervous system disorders) | 51 | 23
Headache (Nervous system disorders) | 104 | 39
Neuropathy peripheral (Nervous system disorders) | 28 | 18
Tremor (Nervous system disorders) | 21 | 5
Adjustment disorder (Psychiatric disorders) | 8 | 9
Alcohol abuse (Psychiatric disorders) | 14 | 15
Anxiety (Psychiatric disorders) | 28 | 21
Depression (Psychiatric disorders) | 26 | 19
Insomnia (Psychiatric disorders) | 87 | 46
Proteinuria (Renal and urinary disorders) | 18 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 28 | 14
Rash (Skin and subcutaneous tissue disorders) | 27 | 9

LIMITATIONS AND CAVEATS:
The primary endpoint was established at 6 months. Treatment, intensive data collection, and statistical power calculations focused on the first 6 months. Given the unexpected placebo + OBR response, cautiously interpret 18, 24, and 30 month outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less